CLINICAL TRIAL: NCT02324504
Title: Evaluation of Electrocardiographic Guidance in Accurate Peripherally Inserted Central Catheter Placement in Children.
Acronym: ECG-PICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Michael Agus, Principal Investigator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00015242
Record Dates: First submitted 2014-11-20; First posted 2014-12-24 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Venous Insufficiency
Keywords: Peripherally Inserted Central Catheter (PICC); Electrocardiographic guidance; Reposition
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placement with C3 Wave Tip System (Experimental): Subjects will have their central catheters placed with the addition of the FDA approved C3 Wave ECG-Based PICC Tip Confirmation System to the standard institution protocol. The system will assist with location of the catheter tip in real-time, during the procedure.
  Interventions: Device: C3 Wave ECG-based PICC Tip Confirmation System

INTERVENTIONS:
Device: C3 Wave ECG-based PICC Tip Confirmation System — The C3 Wave PICC tip detection system will be used to identify catheter tip location during the procedural placement of the catheter. This system includes an ECG monitor that will be connected to the guidewire used for catheter placement. The changes in the ECG tracing will guide correct catheter placement.

SUMMARY:
This study will enroll up to 192 children less than 18 years of age, who will receive electrocardiographic guidance for placement of a PICC in addition to radiography done as standard care. The investigators will determine the location of the PICC tip from both ECG and radiograph, and then measure the degree of correlation between the two methods.

DETAILED DESCRIPTION:
The placement of peripherally inserted central catheters (PICCs) is an important component of medical care for a variety of patients. Current practice requires radiographic confirmation of catheter tip placement prior to use of the line for administration of medications. Often the final catheter tip position may be uncertain based on radiographic imaging. Other times, the catheter is malpositioned and requires adjustment and repeat radiographic imaging. In adult patients, a system of confirmation that is based on electrocardiographic activity has been implemented and is FDA approved. This study will enroll up to 192 children less than 18 years of age who will receive electrocardiographic guidance for placement of a PICC, in addition to radiography done as standard care. The investigators will determine the location of the PICC tip from both ECG and radiograph, and then measure the degree of correlation between the two methods.

ELIGIBILITY:
Inclusion Criteria:

* Age from birth to 17 years in need of a PICC as part of the medical treatment plan
* Suitable for an upper extremity PICC placement
* Hemodynamically stable, including patients stable on vasopressors

Exclusion Criteria:

* Hemodynamic instability
* Cardiac abnormality which leads to abnormal p-wave on ECG
* Arrhythmia at baseline, documented duirng the current hospital admission
* Presence of pacemaker or pacing wires which are currently actively pacing
* Patients who have undergone reconstructive cardiac surgery and/or have anatomic variance that would affect the location of the sinoatrial node in relation to the superior vena cava
* Premature neonate (<37 weeks estimated gestational age)
* Placement of PICC in lower extremity

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael SD Agus, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share with investigators based upon specific requests.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in January 2016 and ended in December 2016. All subjects received the study intervention at Boston Children's Hospital (Boston, MA).
Pre-assignment Details: Participants (or appropriate parent/guardian) gave consent prior to placement of the peripherally inserted central catheter (PICC).
Groups:
- Intervention: Subjects will have their central catheters placed with the assistance of the FDA approved C3 Wave PICC Tip Confirmation System which will assist with location of the catheter tip in real-time, during the procedure.
  C3 Wave ECG-based PICC Tip Confirmation System: The C3 Wave PICC tip detection system will be used to identify catheter tip location during the procedural placement of the catheter. This system includes an ECG monitor that will connected to the guidewire used for catheter placement. The changes in the ECG tracing will guide correct catheter placement. Standard care chest radiograph will be performed as a second measure to confirm catheter tip placement.
Period: Overall Study
Arm/Group | Intervention
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Subjects will have their central catheters placed with the assistance of the FDA approved C3 Wave PICC Tip Confirmation System which will assist with location of the catheter tip in real-time, during the procedure.
  C3 Wave ECG-based PICC Tip Confirmation System: The C3 Wave PICC tip detection system will be used to identify catheter tip location during the procedural placement of the catheter. This system includes an ECG monitor that will be connected to the guidewire used for catheter placement. The changes in the ECG tracing will guide correct catheter placement.
  Chest radiograph: Chest radiograph will be performed as a second measure to confirm catheter tip placement.
Arm/Group | Intervention
Number analyzed (Participants) | 60
Age, Customized [Count of Participants; unit: Participants]
  0-2 Years | 23
  3-11 Years | 14
  12-17 Years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Placement of Peripherally Inserted Central Catheter (PICC)
Description: Successful placement (based upon review of chest radiograph) of the PICC as determined by the tip location of:
  * RA SVC junction (right atrium/superior vena cava) or
  * Distal or lower SVC
Time Frame: Less than 24 hours
Measure: Count of Participants; unit: Participants
Groups:
- Total Enrolllment: All subjects (less than 18 years of age) will have PICC placement guided by the C3 Wave device in order to determine if success rates, overall and by age group, are greater than local historical success rates.
- Subjects Age 0-2 Years of Age: Approximately 38% of the enrolled subjects were two years of age or younger. In all three groups PICC placement will be guided by the C3 Wave device in order to determine if success rates, overall and by age group, are greater than local historical success rates.
- Subjects Age 3-11 Years of Age: Approximately 23% of the enrolled subjects were between the ages of 3 and 11 years. In all three groups PICC placement will be guided by the C3 Wave device in order to determine if success rates, overall and by age group, are greater than local historical success rates.
- Subjects Age 12-17 Years of Age: Approximately 38% of the enrolled subjects were between 12 and 17 years of age. In all three groups PICC placement will be guided by the C3 Wave device in order to determine if success rates, overall and by age group, are greater than local historical success rates.
Arm/Group | Total Enrolllment | Subjects Age 0-2 Years of Age | Subjects Age 3-11 Years of Age | Subjects Age 12-17 Years of Age
Number analyzed (Participants) | 60 | 23 | 14 | 23
Participants | 40 | 14 | 8 | 18

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events from the time of placement of the first electrode until confirmation of the PICC tip location via chest radiography or echocardiography, assessed up to 72 hours.
Groups:
- Intervention: Subjects will have their central catheters placed with the assistance of the FDA approved C3 Wave PICC Tip Confirmation System which will assist with location of the catheter tip in real-time, during the procedure.
  C3 Wave ECG-based PICC Tip Confirmation System: The C3 Wave PICC tip detection system will be used to identify catheter tip location during the procedural placement of the catheter. This system includes an ECG monitor that will connected to the guidewire used for catheter placement. The changes in the ECG tracing will guide correct catheter placement.
  Chest radiograph: Chest radiograph will be performed as a second measure to confirm catheter tip placement.
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No